CLINICAL TRIAL: NCT05820048
Title: The Efficacy and Safety of Proton Pump Inhibitor ( in Patients With Moderate Bleeding Risk and Coronary Artery Disease Undergoing Percutaneous Coronary: A Randomised, Open ,Compared With Control
Brief Title: The Efficacy and Safty of Proton Pump Inhibitor (Lansoprazole)
Acronym: PPI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Daejeon St. Mary's hospital (Other)
Collaborators: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Kim Dae-Won, assistant professor, Daejeon St. Mary's hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DWKim
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Coronary Artery Disease
Keywords: proton pump inhibitor; percutaneous coronary intervention; gastrointestinal bleeding of moderate risk; dual anti-platelet drugs
MeSH Terms: conditions — Coronary Artery Disease | interventions — Lansoprazole

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- proton pump inhibitor (Active Comparator): 1. medication : Lanston
  2. capacity : 15mg
  3. Number of times : QD
  4. period : 6 month
  5. Injection path : oral
  Interventions: Drug: Lansoprazole 15 mg
- non-administered army (No Intervention): No Intervention

INTERVENTIONS:
Drug: Lansoprazole 15 mg — 1. Short-term treatment of active duodenal ulcer
  2. Short-term treatment of active benign gastric ulcers
  3. Thin heat of Helicobacter pylori to prevent recurrence of duodenal ulcer
  4. Maintain duodenal ulcer after treatmentLaw
  5. Treatment of nonsteroidal anti-inflammatory analgesics-induced gastric ulcers
  6. Reducing the risk of developing nonsteroidal anti-inflammatory analgesic-induced gastric ulcers
  7. Short-term treatment of gastroesophageal reflux disease
  8. Short-term treatment of erosive reflux esophagitis
  9. Post-treatment maintenance therapy for erosive reflux esophagitis
  10. Pathological hyperdivision, including Zolinger Ellison syndrome
  Other Names: non-administered army
  Arms: proton pump inhibitor

SUMMARY:
Among patients who performed percutaneous coronary intervention (PCI) in patients with coronary artery disease (CAD), enrollment is performed in patients with moderate risk in gastrointestinal risk assessment indicators. After obtaining the consent form, patients are randomly assigned to the gastric acid secretion inhibitor group and the non-dose group.

Researchers and subjects proceed with the treatment group assignment, treatment-group assignment uses a random number table and the assigned drug is disclosed. Random checks are generated by statisticians and managed by the researchers.

In the test group, the incidence of gastrointestinal clinical events in DAPT patients is expected to be low while taking PPI, but there is a burden of PPI costs. In the case of the control group, the burden of PPI costs is reduced, but there is a possibility that the incidence of clinical events may occur, although it is a small number. Subjects in the test group will take DAPT for at least 6 months from the time of registration, and NSAIDs drugs or steroids and NOAC or warfarin should be prohibited as combination taboo drugs when participating in the study. Data will be collected during normal medical procedures and will be checked through an endoscope in case of upper gastrointestinal bleeding

DETAILED DESCRIPTION:
1. Purpose : This study compares gastrointestinal and cardiovascular events with coronary artery disease (CAD) patients who underwent percutaneous coronary angioplasty in patients with moderate gastrointestinal bleeding risk with use of dual antiplatelet drugs (DAPT), especially controversial use of prophylactic acid secretion inhibitors, and attempts to confirm the effectiveness and safety of gastric acid secretion inhibitors
2. Background : DPAT is a standard treatment in patients with CAD with percutaneous coronary intervention (PCI). However, it is important to consider the GI bleeding risk when using DAPT and to determine whether Proton Pump Inhibitor (PPI) should be prescribed to prevent such accidents. DAPT, or aspirin and P2Y12 receptor inhibitor, complementarily reduce platelet activation and aggregation and consequently reduce the progression of coronary thrombosis.

   We have reported whether PPI use is associated with ischemic events or mortality in patients with DAPT up to date, but we have shown conflicting results depending on the type of study conducted. Observational studies generally show that PPI increases all-cause and cardiovascular mortality, angina and stroke, while RCT studies show that it does not. This difference can be explained by the selection bias. This is because observational studies attempt to reduce selective bias through correction of basic patient characteristics, but unmeasured differences in underlying variables continue to affect the results.
3. method : Among patients who performed PCI in patients with CAD, enrollment is performed in patients with moderate risk in gastrointestinal risk assessment indicators. After obtaining the consent form, patients are randomly assigned to the gastric acid secretion inhibitor group and the non-dose group.

Researchers and subjects proceed with the treatment group assignment, treatment-group assignment uses a random number table and the assigned drug is disclosed. Random checks are generated by statisticians and managed by the researchers.

In the test group, the incidence of gastrointestinal clinical events in DAPT patients is expected to be low while taking PPI, but there is a burden of PPI costs. In the case of the control group, the burden of PPI costs is reduced, but there is a possibility that the incidence of clinical events may occur, although it is a small number. Subjects in the test group will take DAPT for at least 6 months from the time of registration, and NSAIDs drugs or steroids and NOAC or warfarin should be prohibited as combination taboo drugs when participating in the study. Data will be collected during normal medical procedures and will be checked through an endoscope in case of upper gastrointestinal bleeding

ELIGIBILITY:
Inclusion Criteria:

* 19 years of age or older
* Coronary artery disease has one or more of the following
* Stable angina
* unstable angina
* N on ST elevation myocardial infarction
* ST elevation myocardial infarction
* Those who are scheduled to receive or are taking dual antiplatelet therapy including aspirin after PCI trials
* A person whose risk of bleeding falls under an intermediate risk group.

Exclusion Criteria:

* age < 19 years
* known allergy to aspirin and clopidogrel
* A person classified as a high-risk group according to the gastrointestinal risk assessment index
* liver cirrhosis
* known iron deficiency anemia
* recent fibrinolytic therapy
* active cancer
* end-stage renal failure
* life expectancy < 1 year
* co-prescription of NSAIDs, corticosteroid and anticoagulant such as NOAC or warfarin
* pregnancy
* mentally or cognitively disabled people
* mechanical ventilation with endotracheal intubation
* Persons who do not agree to participate in the study
* persons related unequally to investigators (students and employees)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of upper gastrointestinal clinical complex | 6 month after randomization
  Upper gastrointestinal bleeding with clear origin,upper gastrointestinal bleeding with unclear origin, potential upper gastrointestinal bleeding or perforation

SECONDARY OUTCOMES:
The occurrence of a cardiovascular clinical complex | 6 month after randomization
  Combined variables of cardiovascular death, non-fatal myocardial infarction, coronary artery reopening, or ischemic stroke

CONTACTS AND LOCATIONS:
Overall Officials: DaeWon Kim, Principal Investigator — Cardiovascular Center, Mary's Hospital,64, Daeheung-ro, Jung-gu, Daejeon, Republic of Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Capodanno D, Alfonso F, Levine GN, Valgimigli M, Angiolillo DJ. ACC/AHA Versus ESC Guidelines on Dual Antiplatelet Therapy: JACC Guideline Comparison. J Am Coll Cardiol. 2018 Dec 11;72(23 Pt A):2915-2931. doi: 10.1016/j.jacc.2018.09.057. PMID 30522654
- [Result] Franchi F, Angiolillo DJ. Novel antiplatelet agents in acute coronary syndrome. Nat Rev Cardiol. 2015 Jan;12(1):30-47. doi: 10.1038/nrcardio.2014.156. Epub 2014 Oct 7. PMID 25286881
- [Result] Abraham NS, Hlatky MA, Antman EM, Bhatt DL, Bjorkman DJ, Clark CB, Furberg CD, Johnson DA, Kahi CJ, Laine L, Mahaffey KW, Quigley EM, Scheiman J, Sperling LS, Tomaselli GF; ACCF/ACG/AHA. ACCF/ACG/AHA 2010 expert consensus document on the concomitant use of proton pump inhibitors and thienopyridines: a focused update of the ACCF/ACG/AHA 2008 expert consensus document on reducing the gastrointestinal risks of antiplatelet therapy and NSAID use. A Report of the American College of Cardiology Foundation Task Force on Expert Consensus Documents. J Am Coll Cardiol. 2010 Dec 7;56(24):2051-66. doi: 10.1016/j.jacc.2010.09.010. No abstract available. PMID 21126648
- [Result] Sabatine MS, Cannon CP, Gibson CM, Lopez-Sendon JL, Montalescot G, Theroux P, Claeys MJ, Cools F, Hill KA, Skene AM, McCabe CH, Braunwald E; CLARITY-TIMI 28 Investigators. Addition of clopidogrel to aspirin and fibrinolytic therapy for myocardial infarction with ST-segment elevation. N Engl J Med. 2005 Mar 24;352(12):1179-89. doi: 10.1056/NEJMoa050522. Epub 2005 Mar 9. PMID 15758000
- [Result] Yusuf S, Zhao F, Mehta SR, Chrolavicius S, Tognoni G, Fox KK; Clopidogrel in Unstable Angina to Prevent Recurrent Events Trial Investigators. Effects of clopidogrel in addition to aspirin in patients with acute coronary syndromes without ST-segment elevation. N Engl J Med. 2001 Aug 16;345(7):494-502. doi: 10.1056/NEJMoa010746. PMID 11519503
- [Result] Moukarbel GV, Bhatt DL. Antiplatelet therapy and proton pump inhibition: clinician update. Circulation. 2012 Jan 17;125(2):375-80. doi: 10.1161/CIRCULATIONAHA.111.019745. No abstract available. PMID 22249527
- [Result] Laine L, Yang H, Chang SC, Datto C. Trends for incidence of hospitalization and death due to GI complications in the United States from 2001 to 2009. Am J Gastroenterol. 2012 Aug;107(8):1190-5; quiz 1196. doi: 10.1038/ajg.2012.168. Epub 2012 Jun 12. PMID 22688850
- [Result] Bhatt DL, Cryer BL, Contant CF, Cohen M, Lanas A, Schnitzer TJ, Shook TL, Lapuerta P, Goldsmith MA, Laine L, Scirica BM, Murphy SA, Cannon CP; COGENT Investigators. Clopidogrel with or without omeprazole in coronary artery disease. N Engl J Med. 2010 Nov 11;363(20):1909-17. doi: 10.1056/NEJMoa1007964. Epub 2010 Oct 6. PMID 20925534
- [Result] Sehested TSG, Carlson N, Hansen PW, Gerds TA, Charlot MG, Torp-Pedersen C, Kober L, Gislason GH, Hlatky MA, Fosbol EL. Reduced risk of gastrointestinal bleeding associated with proton pump inhibitor therapy in patients treated with dual antiplatelet therapy after myocardial infarction. Eur Heart J. 2019 Jun 21;40(24):1963-1970. doi: 10.1093/eurheartj/ehz104. PMID 30851041
- [Result] Schoenfeld AJ, Grady D. Adverse Effects Associated With Proton Pump Inhibitors. JAMA Intern Med. 2016 Feb;176(2):172-4. doi: 10.1001/jamainternmed.2015.7927. No abstract available. PMID 26751904
- [Result] Moayyedi P, Eikelboom JW, Bosch J, Connolly SJ, Dyal L, Shestakovska O, Leong D, Anand SS, Stork S, Branch KRH, Bhatt DL, Verhamme PB, O'Donnell M, Maggioni AP, Lonn EM, Piegas LS, Ertl G, Keltai M, Bruns NC, Muehlhofer E, Dagenais GR, Kim JH, Hori M, Steg PG, Hart RG, Diaz R, Alings M, Widimsky P, Avezum A, Probstfield J, Zhu J, Liang Y, Lopez-Jaramillo P, Kakkar AK, Parkhomenko AN, Ryden L, Pogosova N, Dans AL, Lanas F, Commerford PJ, Torp-Pedersen C, Guzik TJ, Vinereanu D, Tonkin AM, Lewis BS, Felix C, Yusoff K, Metsarinne KP, Fox KAA, Yusuf S; COMPASS Investigators. Safety of Proton Pump Inhibitors Based on a Large, Multi-Year, Randomized Trial of Patients Receiving Rivaroxaban or Aspirin. Gastroenterology. 2019 Sep;157(3):682-691.e2. doi: 10.1053/j.gastro.2019.05.056. Epub 2019 May 29. PMID 31152740
- [Result] Valgimigli M, Bueno H, Byrne RA, Collet JP, Costa F, Jeppsson A, Juni P, Kastrati A, Kolh P, Mauri L, Montalescot G, Neumann FJ, Petricevic M, Roffi M, Steg PG, Windecker S, Zamorano JL, Levine GN; ESC Scientific Document Group; ESC Committee for Practice Guidelines (CPG); ESC National Cardiac Societies. 2017 ESC focused update on dual antiplatelet therapy in coronary artery disease developed in collaboration with EACTS: The Task Force for dual antiplatelet therapy in coronary artery disease of the European Society of Cardiology (ESC) and of the European Association for Cardio-Thoracic Surgery (EACTS). Eur Heart J. 2018 Jan 14;39(3):213-260. doi: 10.1093/eurheartj/ehx419. No abstract available. PMID 28886622
- See also: ACC/AHA Versus ESC Guidelines on Dual Antiplatelet Therapy: JACC Guideline Comparison — https://pubmed.ncbi.nlm.nih.gov/30522654/
- See also: Novel antiplatelet agents in acute coronary syndrome — https://pubmed.ncbi.nlm.nih.gov/25286881/
- See also: ACCF/ACG/AHA 2010 expert consensus document on the concomitant use of proton pump inhibitors and thienopyridines: a focused update of the ACCF/ACG/AHA 2008 expert consensus document on reducing the gastrointestinal risks of antiplatelet therapy and NSAID — https://pubmed.ncbi.nlm.nih.gov/21126648/
- See also: Addition of clopidogrel to aspirin and fibrinolytic therapy for myocardial infarction with ST-segment elevation — http://pubmed.ncbi.nlm.nih.gov/15758000/
- See also: Effects of clopidogrel in addition to aspirin in patients with acute coronary syndromes without ST-segment elevation — http://pubmed.ncbi.nlm.nih.gov/11519503/
- See also: Antiplatelet therapy and proton pump inhibition: clinician update — https://pubmed.ncbi.nlm.nih.gov/22249527/
- See also: Trends for incidence of hospitalization and death due to GI complications in the United States from 2001 to 2009 — https://pubmed.ncbi.nlm.nih.gov/22688850/
- See also: Clopidogrel with or without omeprazole in coronary artery disease — https://pubmed.ncbi.nlm.nih.gov/20925534/
- See also: Reduced risk of gastrointestinal bleeding associated with proton pump inhibitor therapy in patients treated with dual antiplatelet therapy after myocardial infarction — https://pubmed.ncbi.nlm.nih.gov/30851041/
- See also: Adverse Effects Associated With Proton Pump Inhibitors — https://pubmed.ncbi.nlm.nih.gov/26751904/
- See also: Safety of Proton Pump Inhibitors Based on a Large, Multi-Year, Randomized Trial of Patients Receiving Rivaroxaban or Aspirin — https://pubmed.ncbi.nlm.nih.gov/31152740/
- See also: 2017 ESC focused update on dual antiplatelet therapy in coronary artery disease developed in collaboration with EACTS: The Task Force for dual antiplatelet therapy in coronary artery disease of the European Society of Cardiology (ESC) and of the European — https://pubmed.ncbi.nlm.nih.gov/28886622/